CLINICAL TRIAL: NCT05833243
Title: Effectiveness of Modified Diaphragmatic Training for Improving GERD-Q Score, Diaphragmatic Excursion, Maximum Inspiratory Pressure and Lung Function in Adults With Gastroesophageal Reflux Disease After Covid-19
Brief Title: Effectiveness of Modified Diaphragmatic Training for Gastroesophageal Reflux Disease Post Covid-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Siti Chandra Widjanantie, Principal Investigator, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 22-11-1417
Record Dates: First submitted 2023-04-25; First posted 2023-04-27 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: GERD; Post COVID-19 Condition; Diaphragm Issues
Keywords: Diaphragmatic Training; GERD-Q Score; Diaphragmatic Excursion; Maximal Inspiratory Pressure; Lung Function; GERD After COVID-19
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Intervention Model Description: Intervention Group (modified diaphragmatic training) and control group (standard diaphragmatic training)
Who Masked: Investigator
Masking Description: single-blinded, only the investigator was blinded, using a randomization center for concealment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional Group (Experimental): Baseline measurement will be done in the rehabilitation center. Participants will receive modified diaphragmatic training using modified diaphragmatic training with increased load every week for strength training (60% from inspiratory muscle strength).
  Weekly follow-up will be taken to reassure the respiratory muscle strength. Prescription for intervention will be determined based on the result of baseline measurement.
  After 4 weeks post-intervention measurement will be taken.
  Interventions: Other: modified diaphragmatic training
- Control Group (Active Comparator): Baseline measurement will be done in the rehabilitation center. Participants will receive standard diaphragmatic training using a sitting position.
  Weekly follow-ups will be taken to remeasure the respiratory muscle strength and training procedure.
  After 4 weeks post-intervention measurements will be taken.
  Interventions: Other: standard diaphragmatic training

INTERVENTIONS:
Other: modified diaphragmatic training — Modified diaphragmatic strength training prescriptions will be given based on the result of baseline assessment. The intensity is 60% from the maximum respiratory muscle strength from baseline and weekly remeasurement. Participants are asked to come for weekly follow-up and commit to do at least 20 sessions of exercise. The training is under supervision of physical medicine and rehabilitation specialist.
  Arms: Interventional Group
Other: standard diaphragmatic training — standard diaphragmatic strength training prescriptions will be given as daily routine, 3 times a day.
  Participants are asked to come for weekly follow-up and commit to do at least 20 sessions of exercise. The training is under supervision of physical medicine and rehabilitation specialist.
  Arms: Control Group

SUMMARY:
The study titled "Effectiveness of Modified Diaphragmatic Training for Improving GERD-Q Score, Diaphragmatic Excursion, Maximum Inspiratory Pressure and Lung Function in Adults With Gastroesophageal Reflux Disease After Covid-19: a Single-blinded Randomized Control Trial" is a clinical trial that aimed to investigate the effectiveness of 4 weeks modified diaphragmatic training (MDT) compare with standard diaphragmatic training for improving GERD-Q score, diaphragmatic excursion, maximum inspiratory pressure, and lung function in adults with gastroesophageal reflux disease (GERD) after COVID-19. The trial was single-blinded and randomized, and it included a total of 50 participants. The results of the study showed that MDT was effective in improving GERD-Q score, diaphragmatic excursion, maximum inspiratory pressure, and lung function in adults with GERD after COVID-19.

DETAILED DESCRIPTION:
The study aims to investigate the effectiveness of modified diaphragmatic training compared with standard diaphragmatic training in adults with gastroesophageal reflux disease after covid-19. The design is a single-center in a national respiratory referral center in Indonesia, single-blinded randomized control trial. A central randomization center used computer-generated tables to allocate treatments. The study will involve a randomized controlled trial with a sample size of 50 adult patients with GERD after covid-19. Participants will be randomly assigned to either a modified diaphragmatic training group or a control group.

Four weeks of training with diaphragmatic training followed by modified diaphragmatic training (MDT) or standard diaphragmatic training. Follow-up 30 days

ELIGIBILITY:
Inclusion Criteria:

* Male and female after recover from moderate COVID-19.
* Six month post COVID-19
* Age 18 to 60 years old
* GERD-Q Score more than 7
* Agree to participate in the study
* Well understanding of the study procedure.

Exclusion Criteria:

* History of ventilator used while COVID
* History of uncontrolled cardiac problems and chronic pulmonary
* Pregnancy or lactation
* History of surgery in the abdomen of the thoracic area
* Severe scoliosis or Kyphotic
* HIV/ AIDS, Autoimmune
* Prolonged use of dyslipidemia drug more than 1 year
* Prolonged use of prokinetic gastric drug more than 4 weeks

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2023-02-08 (Actual); Primary Completion 2023-04-14 (Actual); Study Completion 2023-04-18 (Actual)

PRIMARY OUTCOMES:
Change from baseline of GERD-Q Score after 4 weeks | base line and week 4
  GERD was diagnosed when the GERD-Q score is above or equal with 8
Change from baseline of Diaphragmatic Excursion after 4 weeks | base line and week 4
  The increase of diaphragm range of movement during inspiration and expiration
Change from baseline of Maximal Inspiratory Pressure after 4 weeks | base line and week 4
  The maximal pressure of inspiratory muscle strength that related to diaphragm strength

SECONDARY OUTCOMES:
Change from baseline of Lung function (FEV1, FVC and ratio FEV1/FVC) after 4 weeks | base line and week 4
  the improvement of FEV1, FVC and ratio FEV1/FVC

CONTACTS AND LOCATIONS:
Overall Officials: Siti C Widjanantie, MD, Principal Investigator — Fakultas Kedokteran Universitas Indonesia
Locations (1):
- Faculty of Medicine, Universitas Indonesia, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Yes
Study Protocol and Study Outcome
Supporting Information: Study Protocol
Time Frame: 4 weeks
Access Criteria: by request to my email: sitichandraw@gmail.com

REFERENCES:
- [Background] Kader M, Hossain MA, Reddy V, Perera NKP, Rashid M. Effects of short-term breathing exercises on respiratory recovery in patients with COVID-19: a quasi-experimental study. BMC Sports Sci Med Rehabil. 2022 Apr 5;14(1):60. doi: 10.1186/s13102-022-00451-z. PMID 35382885
- [Background] Saha S, Sharma K. Modification of Lifestyle to Recover from Post-COVID Symptoms: A Short Review. J Lifestyle Med. 2022 Sep 30;12(3):113-118. doi: 10.15280/jlm.2022.12.3.113. PMID 36628181
- [Background] Qiu K, Wang J, Chen B, Wang H, Ma C. The effect of breathing exercises on patients with GERD: a meta-analysis. Ann Palliat Med. 2020 Mar;9(2):405-413. doi: 10.21037/apm.2020.02.35. Epub 2020 Mar 17. PMID 32233626